CLINICAL TRIAL: NCT06619418
Title: Assessment of Usability and Satisfaction With a Take-home Device Presenting Sound and Body Stimulation for Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: ENT-2024-33112
Record Dates: First submitted 2024-07-17; First posted 2024-10-01 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Chronic Lower Back Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- device group (Experimental)
  Interventions: Device: TENS device
- Integrative health modality group (Active Comparator)
  Interventions: Behavioral: Integrative health modalities

INTERVENTIONS:
Device: TENS device — will be using an FDA- cleared TENS device for electrical stimulation (TENS 7000, Compass Health Brands) in combination with commercially-available headphones for acoustic stimulation (AKG 845 BT).Will be shown how to use the device, trained on the multimodal stimulation procedure, and sent home with the device for 12 weeks.
  Arms: device group
Behavioral: Integrative health modalities — will be instructed on the integrative health modalities for this study. They will be given a tablet that includes the videos for the visually guided deep breathing. They will also receive the reflective journal and be set up for health coaching visits. At the end of the 12 weeks, this group of participants will return to the U of M campus and complete an interview about satisfaction and usability of the IH modalities.
  Arms: Integrative health modality group

SUMMARY:
Pain symptoms can have a variety of ways to be treated, from medications to physical therapy, with several options being available to patients. However, no one treatment may work for all people who experience pain, especially cLBP. The purpose of this study is to measure the compliance, usability, and satisfaction of an at-home, multi-modal stimulation device in a diverse population of people with chronic lower back pain (cLBP). The multi-modal device will include a combination of electrical stimulation, auditory stimulation, and integrative-health techniques, including mindfulness breathing, health coaching, and reflective journaling. The multi-modal device creation is based on prior knowledge in lower back pain treatment, which includes electrical stimulation of the back (Transcutaneous Electrical Nerve Stimulator or TENS) and integrative health modalities. In isolation, these treatments are only somewhat effective in reducing symptoms.

This pilot study will involve participants who experience cLBP as we investigate a novel at-home, multi-modal device design. The main objective of the pilot usability study is to examine compliance to the intended use of the multi-modal device and approach, as well as protocol feasibility, and satisfaction with the settings and design.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older
* Must be within commuting distance to the University of Minnesota
* Able to provide consent and follow study instructions
* Must be able to understand English
* Must have chronic LBP, which is defined as lower back pain for more than 3 months
* A score of 4 or higher on the PEG
* Must be willing to commit to full duration of the study
* Not currently taking any benzodiazepines or sedative hypnotics

Exclusion Criteria:

* Back Pain associated with:
* Spondylolisthesis or spinal stenosis
* Sciatica or radiculopathy
* Rhematologic or inflammatory disease
* Trauma, fracture, dislocation, or previous back surgery
* A score of 10 on the PEG
* Pregnant
* Have an electrically implanted device, such as a pacemaker.
* Heart Disease
* Epilepsy
* Cancer
* Psychiatric conditions including psychosis, suicidal ideation, or substance abuse disorder
* A pure tone average of more than 40 dB HL at 500 dB, 1000 dB, or 2000 dB HL.
* Individuals currently using other lower back pain treatments during the study in which they are unable to maintain a steady state while participating in our study for one month before beginning the multi-modal regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-08-11 (Estimated); Study Completion 2026-08-11 (Estimated)

PRIMARY OUTCOMES:
compliance rate | 12 weeks
  Measure compliance in terms of time using the integrative health devices and the multi-modal stimulation device over a period of 12 weeks to determine the effect on participant compliance by adding electrical stimulation to the device.

SECONDARY OUTCOMES:
satisfaction rate | 12 weeks
  relating to usability of an at-home multi-modal stimulation approach and device and integrative health practices..

CONTACTS AND LOCATIONS:
Overall Officials: Molly Sturges, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States